CLINICAL TRIAL: NCT07193264
Title: CaffeineHSC - Effect of Chronic Caffeine Consumption and Acute Caffeine Administration on the Hematopoietic System
Brief Title: Impact of Chronic and Acute Caffeine Intake on the Hematopoietic System
Acronym: CaffeineHSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jasmin Rettkowski (Other)
Collaborators: ETH Zurich (Other); Laboratory of Stem Cell Biology and Ageing, ETH Zurich, Prof. Nina Cabezas-Wallscheid (Unknown); Prof. Dr. Nina Cabezas-Wallscheid, ETH Zurich (Unknown)
Responsible Party: Sponsor-Investigator, Jasmin Rettkowski, Dr. Jasmin Rettkowski, Principal Investigator, Department of Health Sciences and Technology, ETH Zurich, ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-00914
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults; Hematopoietic System; Caffeine
Keywords: Caffeine consumption; caffeine; Hematopoietic Stem Cells; Hematopoietic Stem and Progenitor Cells; Effect of caffeine on blood system; Effect of caffeine on hematopoietic system
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: This is a single-group, open-label study in which all participants receive a single oral dose of 200 mg caffeine under fasting conditions. Blood samples are collected before and three hours after caffeine intake to assess mobilization, function, gene expression, and metabolic profile of hematopoietic stem and progenitor cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caffeine intervention (Experimental): 200mg Caffeine
  Interventions: Other: Caffeine (200 mg)

INTERVENTIONS:
Other: Caffeine (200 mg) — Participants receive a single oral dose of 200 mg caffeine under fasting conditions. Blood samples are collected before and three hours after intake to evaluate effects on hematopoietic stem and progenitor cells, including mobilization, function, gene expression, and metabolism.

SUMMARY:
This study investigates how caffeine intake affects blood stem and progenitor cells in healthy adults.

The trial will compare people who regularly consume caffeine with those who consume very little or none. All participants will receive a single 200 mg caffeine tablet (similar to one cup of coffee) under fasting conditions. Blood samples will be collected before and three hours after caffeine intake.

The study will assess whether caffeine influences the mobilization of blood stem and progenitor cells from the bone marrow into the bloodstream. It will also examine the effects of caffeine on the function, gene activity, and metabolism of blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Able to give consent.
* Healthy adults aged ≥ 18 years.
* Regular caffeine consumers (≥1 coffee cup/day or ≥1 energy drink/day) or non-consumers (≤1 cup/month and ≤1 energy drink/month) for at least 6 months.
* Willingness to comply with fasting requirements and study procedures.

Exclusion Criteria:

* Chronic illnesses or medication use affecting metabolism, including metabolic disorders (e.g., diabetes, thyroid dysfunction, metabolic syndrome).
* Personal history of cancer.
* Personal history of hematological disorders.
* History of radiation therapy.
* Known caffeine hypersensitivity or intolerance.
* Known immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mobilization of hematopoietic stem and progenitor cells | From baseline to three hours after caffeine intake
  The change in the numbers of mobilized HSPCs (defined as CD34+ cells) [cells/ml] in blood (measured by flow cytometry) from baseline to three hours after intake of a single oral dose of 200mg caffeine in habitual caffeine consumers versus non-caffeine consumers.
Mobilization of hematopoietic stem and progenitor cells | From baseline to three hours after caffeine intake
  The change in the relative abundance of HSPCs [% HSPCs of total PBMCs] in blood (measured by flow cytometry) from baseline to three hours after intake of a single oral dose of 200mg caffeine in habitual caffeine consumers versus non-caffeine consumers.

SECONDARY OUTCOMES:
Functional alterations in CD34+ peripheral blood cells | From baseline to three hours after caffeine intake
  Functional alterations in CD34+ PB cells: self-renewal [number of colonies] assessed via colony-forming unit assay.
Functional alterations in CD34+ peripheral blood cells | From baseline to three hours after caffeine intake
  Functional alterations in CD34+ PB cells: single HSPC proliferation [number of cell divisions within 72h] assessed via single HSC proliferation assay.
Transcriptional changes in CD34+ cells | From baseline to three hours after caffeine intake
  Transcriptional changes in CD34+ cells [log2 fold change in gene expression and DEG count] assessed via single-cell RNA sequencing.
Relative metabolite abundance | From baseline to three hours after caffeine intake
  Relative metabolite abundance [arbitrary units based on peak area or height in LC-MS] in plasma and intracellularly in isolated CD34+ cells.
Change in the numbers of peripheral blood cells | From baseline to three hours after caffeine intake
  The change in the numbers of PB cells [cells/ml], including B cells, T cells, myeloid cells in blood, and relative, and measured by flow cytometry
Change in the numbers of peripheral blood cells | From baseline to three hours after caffeine intake
  The change in relative abundance of PB cells [% cell type of total PBMCs] including B cells, T cells, myeloid cells in blood, and measured by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- ETH GLC, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes